CLINICAL TRIAL: NCT07165873
Title: Comparison of the Analgesic Efficacy of Erector Spinae Plane Block, Serratus Anterior Plane Block, and Serratus Posterior Superior Intercostal Plane Block on Postoperative Pain in Patients Undergoing Video-Assisted Thoracoscopic Surgery
Brief Title: Comparison of ESP, SAP and SPSIP Blocks on VATS'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Oguz Gundogdu, Associate Professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2023-05/04
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain Management
Keywords: erector spinae plane block; serratus anterior plane block; serratus posterior superior intercostal plane block; video-assisted thoracoscopic surgery; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESP block (Active Comparator): Erector spinae plane (ESP) block was performed in 15 patients. An ultrasound (USG) probe was placed in a sagittal orientation at the T5 level, 3 cm lateral to the midline, to visualize the transverse process. The trapezius, rhomboid major, and erector spinae muscles were identified. Using an in-plane technique, a needle was advanced cranio-caudally through these muscles until it reached the transverse process. After negative aspiration, 30 mL of 0.25% bupivacaine was injected deep to the erector spinae muscle. The block was performed unilaterally, targeting the surgical hemithorax.
  Interventions: Procedure: Erector Spinae Plane Block
- SAP block (Active Comparator): Serratus anterior plane (SAP) block was performed in 15 patients. The latissimus dorsi and serratus anterior muscles were identified by using USG at the midaxillary line at the 4th-5th rib level in a longitudinal parasagittal orientation. A needle was advanced from caudal to cranial using an in-plane approach, first targeting the plane between the latissimus dorsi and serratus anterior, and then deep to the serratus anterior. After negative aspiration, 10 mL was injected into the superficial plane and 20 mL into the deep plane, for a total of 30 mL of 0.25% bupivacaine. The block was performed unilaterally, targeting the surgical hemithorax.
  Interventions: Procedure: Serratus anterior plane block (SAP)
- SPSIP block (Active Comparator): The USG probe was placed 2-3 cm medial to the scapular spine to visualize the trapezius, rhomboid major, and serratus posterior superior muscles. At the level of the 2nd-3rd ribs, a needle was advanced into the plane between the serratus posterior superior muscle and the rib. After confirming negative aspiration, 30 mL of 0.25% bupivacaine was injected. The block was performed unilaterally, targeting the surgical hemithorax.
  Interventions: Procedure: Serratus posterior superior intercostal plane block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — 30 mL of 0.25% bupivacaine was injected deep to the erector spinae muscle.
  Other Names: ESP block
  Arms: ESP block
Procedure: Serratus anterior plane block (SAP) — 10 mL was injected into the superficial plane and 20 mL into the deep plane, for a total of 30 mL of 0.25% bupivacaine.
  Other Names: SAP block
  Arms: SAP block
Procedure: Serratus posterior superior intercostal plane block — 30 mL of 0.25% bupivacaine was injected into the plane between the serratus posterior superior muscle and the rib.
  Other Names: spsip block
  Arms: SPSIP block

SUMMARY:
This study aimed to compare erector spinae plane block (ESPB), serratus anterior plane block (SAPB), and serratus posterior superior intercostal plane block (SPSIPB) to determine the most suitable technique for maintaining postoperative analgesia in video-assisted thoracoscopic surgeries (VATS).

DETAILED DESCRIPTION:
Patients were randomly allocated into three groups: ESPB, SAPB, and SPSIPB. All patients received postoperative paracetamol and dexketoprofen, and intravenous tramadol hydrochloride was administered via patient-controlled analgesia. Postoperative static and dynamic VAS scores, total tramadol consumption, side effects, and the need for additional analgesia were monitored and recorded at regular intervals. Primary outcome was VAS scores and secondary outcome was total tramadol consumption.

Block Techniques

All blocks were performed following surgical closure, prior to extubation, with the patient in lateral decubitus and the skin prepared with 10% povidone-iodine.

ESPB was performed in 15 patients. An ultrasound (USG) probe was placed in a sagittal orientation at the T5 level, 3 cm lateral to the midline, to visualize the transverse process. The trapezius, rhomboid major, and erector spinae muscles were identified. Using an in-plane technique, a needle was advanced cranio-caudally through these muscles until it reached the transverse process. After negative aspiration, 30 mL of 0.25% bupivacaine was injected deep to the erector spinae muscle.

SAPB: The latissimus dorsi and serratus anterior muscles were identified at the midaxillary line at the 4th-5th rib level in a longitudinal parasagittal orientation. A needle was advanced from caudal to cranial using an in-plane approach, first targeting the plane between the latissimus dorsi and serratus anterior, and then deep to the serratus anterior. After negative aspiration, 10 mL was injected into the superficial plane and 20 mL into the deep plane, for a total of 30 mL of 0.25% bupivacaine.

SPSIPB: The USG probe was placed 2-3 cm medial to the scapular spine to visualize the trapezius, rhomboid major, and serratus posterior superior muscles. At the level of the 2nd-3rd ribs, a needle was advanced into the plane between the serratus posterior superior muscle and the rib. After confirming negative aspiration, 30 mL of 0.25% bupivacaine was injected.

All blocks were performed unilaterally, targeting the surgical hemithorax.

Postoperative Analgesia and Assessments

Twenty minutes before extubation, all patients received 1 g IV paracetamol and 50 mg IV dexketoprofen. In the recovery room, patient-controlled analgesia (PCA) with IV tramadol hydrochloride was initiated (4 mg/mL concentration, 10 mg bolus, 20-minute lockout, maximum 3 boluses/hour).

Postoperative VAS scores (static at rest and dynamic during movement or coughing) were recorded at 0, 1, 6, 12, 18, and 24 hours. The first VAS assessment (0 hour) was performed when the patient achieved an Aldrete score of 9. If VAS ≥ 4, an additional 1 g IV paracetamol (maximum 3 g/day) was administered. Additional analgesic consumption was recorded. Side effects such as nausea, vomiting, and pruritus were documented.

ELIGIBILITY:
Inclusion Criteria:

* Forty-five adult patients scheduled for elective wedge resection or biopsy under VATS, classified as American Society of Anesthesiologists (ASA) physical status I-III, were enrolled after providing written informed consent.

Exclusion Criteria:

* ASA class IV or higher,
* morbid obesity (BMI > 40 kg/m²),
* body weight ≤ 50 kg,
* skin infection at the block site,
* refusal to participate,
* inability to cooperate during postoperative pain assessment,
* conversion to open surgery,
* preexisting pain,
* known allergy to any study medication,
* coagulopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) score | postoperative 24 hours
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10 cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

SECONDARY OUTCOMES:
Total tramadol consumption | postoperative 24 hours
  Postoperative total analgesic (tramadol) need was recorded as "milligram" in unit.

CONTACTS AND LOCATIONS:
Overall Officials: Oğuz Gündoğdu, Principal Investigator — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No